CLINICAL TRIAL: NCT03019016
Title: A Multi-Center Retrospective Comparison of Intracorporeal and Extracorporeal Anastomoses for Minimally Invasive Right Colectomy
Brief Title: Comparison of Intracorporeal and Extracorporeal Anastomoses for Minimally Invasive Right Colectomy
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-dVRC-001
Record Dates: First submitted 2016-08-29; First posted 2017-01-12 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Colonic Neoplasms; Crohn Disease
MeSH Terms: conditions — Colonic Neoplasms; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Robotic RC (IA): Benign or malignant disease under going a right colectomy.
  Interventions: Procedure: Right Colectomy
- Robotic RC (EA): Patients with benign or malignant disease under going a right colectomy.
  Interventions: Procedure: Right Colectomy
- Laparoscopic RC (IA): Patients with benign or malignant disease under going a right colectomy.
  Interventions: Procedure: Right Colectomy
- Laparoscopic RC (EA): Patients with benign or malignant disease under going a right colectomy.
  Interventions: Procedure: Right Colectomy

INTERVENTIONS:
Procedure: Right Colectomy — Robotic-assisted or laparoscopic right colectomy with intracorporeal or extracorporeal anastomosis either on or proximal to midtransverse colon.

SUMMARY:
The primary objective of this study is to retrospectively compare the perioperative and short-term (discharge through 30 days) outcomes of intracorporeal and extracorporeal anastomosis in minimally invasive right colectomies for benign and malignant disease.

The secondary objective of this study is to retrospectively compare the rates of incisional hernia (up to 6 month post procedure) between intracorporeal and extracorporeal arms.

DETAILED DESCRIPTION:
This is a multi-center, retrospective chart review study of all consecutive cases of right colectomy performed by participating surgeons at their respective institutions that meet all inclusion and exclusion criteria. All cases of right colectomy performed with intracorporeal or extracorporeal anastomoses or via laparoscopic or robotic platforms that meet the study inclusion and exclusion criteria, will be considered for inclusion. The chart review will be performed in a reverse chronological order starting at a minimum of 30 days prior to IRB approval of the study at the site until the number of robotic-assisted and laparoscopic cases to be included per surgeon has been met. Study initiation at the participating site will occur once a research agreement has been executed between Intuitive Surgical and the participating Institution/Investigator and IRB approval has been obtained.

It is anticipated that the retrospective chart review will span the period between January 1, 2010 through 30-days prior to IRB approval of the study in 2016. Baseline patient characteristics, perioperative and post-operative short term clinical and pathological outcomes, and incisional hernia data will be obtained from hospital records for a total of up to approximately 1000 robotic and laparoscopic cases, among the 4 subgroups: robotic-assisted right colectomy with intracorporeal anastomosis (RRCIA), robotic-assisted right colectomy with extracorporeal anastomosis (RRCEA), laparoscopic right colectomy with intracorporeal anastomosis (LRCIA) and laparoscopic right colectomy with extracorporeal anastomosis (RRCEA). Since the data will have been de-identified, and is archival in nature, there will be no active subject recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with benign or malignant right colon disease
* Patients who have undergone robotic-assisted or laparoscopic right colectomy with intracorporeal or extracorporeal anastomosis either on or proximal to mid-transverse colon

Exclusion Criteria:

* Patients with perforated, obstructing or locally invasive neoplasm (T4b)
* Emergency procedures
* Patients undergoing right colectomy as a secondary procedure
* Patients undergoing radiation therapy for malignant neoplasia before and after procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age ≥ 18 years Patients with benign or malignant right colon disease Patients who have undergone robotic-assisted or laparoscopic right colectomy with intracorporeal or extracorporeal anastomosis either on or proximal to mid-transverse colon
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Chart review on PeriOperative Information | Intraoperative through 30-days follow-up
  Number of complications observed intraoperatively through 30-days

SECONDARY OUTCOMES:
Chart review on Postoperative Information | Postoperative through 6 month follow-up
  Number of complications observed postoperatively through 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Shilpa Mehendale, Study Director — Sr Director, Clinical Affairs, Intuitive Surgical, Inc.

IPD SHARING:
Plan to Share IPD: Yes